CLINICAL TRIAL: NCT04290403
Title: A Randomised Cross Over Trial of Briefs With Tapes Versus Pull Ups for the Containment of Urinary Incontinence in Community Dwelling Older People Living With Mild to Moderate Dementia (CUPID)
Brief Title: Briefs With Tapes Versus Pull Ups for Urinary Incontinence in Older People With Mild to Moderate Dementia (CUPID)
Acronym: CUPID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Alberta (Other)
Collaborators: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CUPID-CDMW-1019
Record Dates: First submitted 2019-12-05; First posted 2020-02-28 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Dementia; Randomised Cross Over Trial; continence products
MeSH Terms: conditions — Urinary Incontinence; Dementia

STUDY DESIGN:
Intervention Model Description: Crossover trial of briefs with tapes versus pull ups for the containment of urinary incontinence
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pull ups (Experimental): Pull-up continence products
  Interventions: Device: Pull Ups
- Styled briefs with tapes (Experimental): Styled briefs with tapes
  Interventions: Device: Styled Briefs with tapes

INTERVENTIONS:
Device: Pull Ups — Participants will be asked to wear pull-ups continence products for the duration of four weeks
  Arms: Pull ups
Device: Styled Briefs with tapes — Participants will be asked to wear styled briefs with tapes for the duration of four weeks
  Arms: Styled briefs with tapes

SUMMARY:
Urinary incontinence is a common health problem that significantly affects the quality of life of older people. The risk of urinary incontinence is increased in people living with dementia. Many products aid the management of urinary incontinence, with many people choosing to manage incontinence with containment products. The purpose of this study is to examine and compare two containment products - pull ups and style briefs with tapes, in self-management of urinary incontinence in people living with dementia.

DETAILED DESCRIPTION:
Urinary incontinence is common in later life and the risk of incontinence is increased in people living with dementia (PLWD). For many, incontinence is managed with toileting assistance containment products, regardless of other potential treatments. As toileting becomes more difficult and incontinence more likely, a containment product which mimics normal underwear, which is familiar to the PLWD may be an attractive option to preserve successful toileting and self management of continence with containment products and toileting for as long as possible. This study is designed to explore the relative benefits or disadvantages of containment with either briefs with tapes or pull ups in the self management of continence by containment products and toileting in PLWD.

Primary objective

To examine the benefits and disadvantages of self-management of urinary incontinence by pulls compared to style briefs with tapes in PLWD.

Research Method/Procedures

This study will comprise a three-phase design

A small sample, exploratory study to ascertain the feasibility of recruitment, trial design and conduct and to enable calculation of an effect size for the trial primary outcome including care partner interviews and exploration of qualitative factors in use not captured elsewhere, economic variables and costs.

A crossover study with an interval washout (pre-trial care) period. Each participant will undergo a 3-day assessment of incontinence severity to ensure eligibility and then, in random order, a four-week period of use of one investigational product, a two week return to their usual care (the care methods undertaken prior to trial commencement) and then a four-week period of use of the comparative investigational product.

A post-treatment phase, qualitative semi-structured interview with PLWD and their care partners to discuss the impressions of the use of each investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Able to toilet independently or independently following prompting or instruction to do so.
* Independently mobile, with or without walking aids
* Use of any type of continence produce, for the management of moderate incontinence.
* Moderate incontinence severity as measured by Incontinence Severity (Sandvik) index.
* Availability of care partner willing to co-operate and participate in trail procedures

Exclusion Criteria:

* Need for daily help with dexterity to apply any continence product
* Waist size or body shape which renders any size of either investigational product inapplicable
* PLWD unable to indicate the need to toilet
* PLWD with significant faecal incontinence
* Permanent residence in nursing home or expected to enter nursing home within two months of trail entry
* Presence of any other condition, which, in the opinion of the investigator makes PLWD unable to participate in the necessary trail procedures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Number of Successful Toileting Episodes | 56 days
  Between group change in the proportion of "successful toileting episodes", defined as episodes of independent toileting with pad use and reapplication without leakage, misapplication or failure, between baseline measurement and end of study investigational product.

SECONDARY OUTCOMES:
Number of continence products used | 56 days
  Number of products used in excess of those deemed necessary [2/24h] according to degree of incontinence.
Number of unintentional leakage | 56 days
  Number of unintentionally leaking products due to misapplication, average per 24h over the duration of the study
Number of episodes leading to unintentionally soiled or wet clothing | 56 days
  Difference in number of episodes leading to wet or unintentionally soiled clothing, between investigational products over the duration of the study.
Number of laundry episodes | 56 days
  Differences in number of laundry episodes(either clothes or bed linen) between investigational products over the duration of the study
Number of hours of care partner time | 56 days
  Difference in care partner time in maintaining continence with investigational products and toileting over the duration of the study
Cost of care partner time | 56 days
  Difference in care partner cost (costed at minimum wage per hour) in maintaining continence with investigational products and toileting over the duration of the study
Quality of life at baseline and end of study | 56 days
  Change in quality of life measures between baseline assessment and end of study using Quality of Life Alzheimer Disease (ADQoL) validated questionnaire.
  The ADQoL scores can be calculated based on patient and caregiver reports and can be combined into a single score, with total scores range from 13 to 52, with higher scores indicating better QoL
Zarit burden index | 56 days
  Comparison of change in Zarit burden index between baseline and end of investigational product use compared between products. Zarit burden index consists of 22 items used to calculate a total score that can range between 0 and 88 (88 = more burden)
Number of Care Partners satisfied with treatment | 56 days
  Persons living with dementia and care partner assessment of satisfaction with each investigational product and its use, assessed at the end of each testing period
Number of PLWD satisfied with treatment | 56 days
  Impressions of ease of use and user satisfaction on the part of persons living with dementia and care partner, at the end of each period of investigational product use, assessed by semi-structured interview

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Geriatric Medicine, Clinical Sciences Building, University of Alberta Hosp, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Hilmer SN, Perera V, Mitchell S, Murnion BP, Dent J, Bajorek B, Matthews S, Rolfson DB. The assessment of frailty in older people in acute care. Australas J Ageing. 2009 Dec;28(4):182-8. doi: 10.1111/j.1741-6612.2009.00367.x. PMID 19951339
- [Background] Logsdon, R.G., , Gibbons, L.E., McCurry, S.M., Teri, L., Quality of life in Alzheimer's disease: patient and caregiver reports. Journal of mental health and ageing, 1999. 5: p. 21-25.
- [Background] Volz-Sidiropoulou E, Rings T, Wagg AS, Leistner N, Gauggel S, Kirschner-Hermanns R. Development and initial psychometric properties of the 'ICIQ-Cog': a new assessment tool to measure the disease-related impact and care effort associated with incontinence in cognitively impaired adults. BJU Int. 2018 Aug;122(2):309-316. doi: 10.1111/bju.14186. Epub 2018 Apr 10. PMID 29509292
- [Background] Baker PS, Bodner EV, Allman RM. Measuring life-space mobility in community-dwelling older adults. J Am Geriatr Soc. 2003 Nov;51(11):1610-4. doi: 10.1046/j.1532-5415.2003.51512.x. PMID 14687391
- [Background] Gotoh M, Matsukawa Y, Yoshikawa Y, Funahashi Y, Kato M, Hattori R. Impact of urinary incontinence on the psychological burden of family caregivers. Neurourol Urodyn. 2009;28(6):492-6. doi: 10.1002/nau.20675. PMID 19090589
- [Background] Hérbert, R., Bravo, G., & Préville, M., Reliability, validity, and reference values of the Zarit Burden Interview for assessing informal caregivers of community-dwelling older persons with dementia. Canadian Journal on Aging, 2000. 19: p. 494-507.
- [Background] Lesen E, Bjorholt I, Ingelgard A, Olson FJ. EXPLORATION AND PREFERENTIAL RANKING OF PATIENT BENEFITS OF MEDICAL DEVICES: A NEW AND GENERIC INSTRUMENT FOR HEALTH ECONOMIC ASSESSMENTS. Int J Technol Assess Health Care. 2017 Jan;33(4):463-471. doi: 10.1017/S0266462317000848. Epub 2017 Oct 25. PMID 29065937